CLINICAL TRIAL: NCT02092116
Title: An Open Phase I/IIa Study to Evaluate the Safety and Effect of Therapeutic HIV-1 Immunization Using Vacc-4x + rhuGM-CSF and HIV-1 Reactivation Using Romidepsin on the Viral Reservoir in Virologically Suppressed HIV-1 Infected Adults on cART
Brief Title: Safety and Efficacy of Romidepsin and the Therapeutic Vaccine Vacc-4x for Reduction of the Latent HIV-1 Reservoir
Acronym: REDUC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bionor Immuno AS (Industry)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BPC01-001; 2013-004747-23 (EudraCT Number)
Record Dates: First submitted 2014-03-03; First posted 2014-03-19 (Estimated); Results first posted 2017-03-01 (Actual); Last update posted 2017-03-01 (Actual); Status verified 2017-01

CONDITIONS: HIV I Infection
MeSH Terms: interventions — romidepsin; Vacc-4x; sargramostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part A (Other): Pre-treatment phase of 2-4 weeks (Visit 1- Visit 2a) followed by viral reactivation phase of 3 weeks (Visit 2 to Visit 7) consisting of one cycle of romidepsin infusions at a dosing of 5 mg/m2 on days 0, 7, and 14.
  Post-activation phase of ~9 weeks (Visit 8 to Visit 11) to assess the effect of romidepsin on the size of latent HIV-1 reservoir.
  Interventions: Drug: Romidepsin
- Part B (Other): Pre-treatment phase of 2-4 weeks (Visit 1-Visit 2) followed by a therapeutic HIV-1 immunization phase of 12 weeks (Visit 2 to Visit 7) in which 1.2 mg Vacc-4x was administered together with 0.06 mg rhuGM-CSF at Visits 2, 3, 4, 5, 6 and 7 follow by a follow-up period of 2 weeks (Visit 8).
  A viral reactivation phase of 3 weeks (Visit 9-Visit 11) consisting of one cycle of 3 romidepsin infusions (5 mg/m2) followed by a post-treatment observation phase of ~9 weeks (Visit 12-Visit 13) to assess the effect of the investigational treatment on the size of the latent HIV-1 reservoir.
  A monitored antiretroviral pause of up to 16 weeks (Visit 14-Visit 33).
  Interventions: Drug: Romidepsin; Biological: Vacc-4x; Biological: rhuGM-CSF

INTERVENTIONS:
Drug: Romidepsin — Latency reversing agent
  Other Names: Istodax®
Biological: Vacc-4x — Vacc-4x is a peptide-based HIV immunotherapy administered intradermally. Vacc-4x peptides are reconstituted in sterile water.
  Other Names: A combination of Vacc-10, Vacc-11, Vacc-12 and Vacc-13
  Arms: Part B
Biological: rhuGM-CSF — Granulocyte macrophage colony stimulating factor as a local adjuvant
  Other Names: Leukine®
  Arms: Part B

SUMMARY:
The REDUC trial's objective is to address one of the core issues with the treatment of HIV, which is that some HIV infected cells hide in so-called latent reservoirs. The reservoirs are unaffected by conventional HIV medication and invisible to the immune system. HDACi have the potential to activate these latently infected cells. This will make the HIV infected cells visible to the immune system; the immune response generate by Vacc-4x will be able to attack and eliminate the infected cells.

DETAILED DESCRIPTION:
The study is divide into two parts. In Part A the safety and tolerability of romidepsin will be evaluated and the effect of romidepsin treatment on HIV-1 transcription in HIV-infected patients virologically suppressed on cART will be determined.

In Part B the effect of treatment with Vacc-4x + rhuGM-CSF and romidepsin treatment on the HIV-1 latent reservoir in HIV-infected patients virologically suppressed on cART will be measured.

Six patients will be enrolled for part A and the safety and tolerability profile evaluated before enrolling 20 patients in B.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years
2. Currently receiving cART and having received cART for a minimum of 1 year
3. HIV-1 plasma RNA <50 copies/mL for at least 1 year (excluding viral load blips)
4. CD4 T cell count ≥500 cells/mm3

Exclusion Criteria:

1. CD4 T cell count nadir <200 cells/mm3
2. Previous treatment with an HDACi (Histone deacetylase inhibitor) within the previous 6 months
3. Any evidence of an active AIDS-defining opportunistic infection, active HBV or HCV co-infection, significant cardiac disease, malignancy, transplantation, insulin dependent diabetes mellitus or other protocol defined excluded medical condition
4. Use of any protocol defined contraindicated medication or vaccination
5. Unacceptable values of the hematologic and clinical chemistry parameters as defined in the protocol.
6. Males or females who are unwilling or unable to use protocol defined methods of contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2014-03; Primary Completion 2015-08 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lars Jørgen Østergaard, MD, PhD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Skejby Sygehus, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: No
Participants have not provided informed consent for their anonymized individual data to be made available beyond that described in the patient information sheet.

REFERENCES:
- [Derived] Leth S, Schleimann MH, Nissen SK, Hojen JF, Olesen R, Graversen ME, Jorgensen S, Kjaer AS, Denton PW, Mork A, Sommerfelt MA, Krogsgaard K, Ostergaard L, Rasmussen TA, Tolstrup M, Sogaard OS. Combined effect of Vacc-4x, recombinant human granulocyte macrophage colony-stimulating factor vaccination, and romidepsin on the HIV-1 reservoir (REDUC): a single-arm, phase 1B/2A trial. Lancet HIV. 2016 Oct;3(10):e463-72. doi: 10.1016/S2352-3018(16)30055-8. Epub 2016 Jul 7. PMID 27658863
- [Derived] Sogaard OS, Graversen ME, Leth S, Olesen R, Brinkmann CR, Nissen SK, Kjaer AS, Schleimann MH, Denton PW, Hey-Cunningham WJ, Koelsch KK, Pantaleo G, Krogsgaard K, Sommerfelt M, Fromentin R, Chomont N, Rasmussen TA, Ostergaard L, Tolstrup M. The Depsipeptide Romidepsin Reverses HIV-1 Latency In Vivo. PLoS Pathog. 2015 Sep 17;11(9):e1005142. doi: 10.1371/journal.ppat.1005142. eCollection 2015 Sep. PMID 26379282

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject screened 6 March 2014 and last subject last visit 25 June 2014 for Part A.
  First subject screened 19 May 2014 and last subject last visit 29 May 2015 for Part B.
  One clinical trial site at Aarhus University Hospital, Denmark
Pre-assignment Details: 7 patients were screened and 6 patients were enrolled in Part A. 24 patients were screened and 20 patients were enrolled in Part B.
Period: Overall Study
Arm/Group | Part A | Part B
Started | 6 | 20
Completed | 6 | 16
Not Completed | 0 | 4
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A | Part B | Total
Number analyzed (Participants) | 6 | 20 | 26
Age, Customized [Number; unit: participants]
  >18 years | 6 | 20 | 26
Gender [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 5 | 17 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 6 | 17 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  Denmark | 6 | 20 | 26
Time since HIV diagnosis [Median (Full Range); unit: years] | 13.3 [7.0 to 22.6] | 9.6 [2.6 to 28.7] | 9.85 [2.6 to 28.7]
Time since HIV infection [Median (Full Range); unit: years] — Population: Information was not available for 2 patients in Part A and for 1 patient in Part B.
  years
    number analyzed (Participants) | 4 | 19 | 23
    (all) | 13.5 [10.7 to 23.1] | 10.2 [2.7 to 31.7] | 12.2 [2.7 to 31.7]
Time since ART initiation [Median (Full Range); unit: years] | 10.05 [4.2 to 14.5] | 6.3 [2.4 to 18.1] | 6.9 [2.4 to 18.1]
Latest pre-ART viral load [Median (Full Range); unit: copies/mL] — Population: Pre-ART viral load was not availabel for 2 patrients in Part B.
  copies/mL
    number analyzed (Participants) | 6 | 18 | 24
    (all) | 123300 [1977 to 2450000] | 67024 [3674 to 10000000] | 72597.5 [1977 to 10000000]
Nadir CD4+ T-cell count [Median (Full Range); unit: 10^6 cells/L] | 246.5 [40 to 340] | 280 [60 to 710] | 267.5 [40 to 710]
Mean CD4+ T-cell counts [Median (Full Range); unit: 10^6 cells/L] | 807.5 [570 to 1015] | 669.8 [465 to 1645] | 712.3 [465 to 1645]

OUTCOME MEASURES:

1. Primary Outcome: Part A: Number of Participants With Adverse Events (AE) and Serious Adverse Events (SAE)
Description: Safety and tolerability evaluation as measured by adverse events (AE) and serious adverse events (SAE).
Time Frame: 3 weeks
Measure: Number; unit: participants
Arm/Group | Part A
Number analyzed (Participants) | 6
participants
  Treatment emergent adverse events | 6
  Adverse reactions, grade 1 | 6
  Adverse reactions, grade 2 | 1
  Related to Romidepsin | 6
  Not related | 3

2. Primary Outcome: Part B: Changes From Baseline in HIV-1 Reservoir (Total HIV-1DNA; Integrated HIV-1 DNA in Unfractionated CD4+ T Cells and Replication Competent Provirus.
Description: Total HIV-1 DNA and integrated HIV-1 DNA were analysed by MMRM analysis (copies/10^6 CD4+ T cells). To estimate the frequency of infectious units per 10^6 resting memory CD4+ T cells a quantitative viral outgrowth assay (qVOA) was used.
  Blood samples were obtained at Day 0, Day 105 and Day 161.
Time Frame: Day 161/175
Population: 4 patients were excluded; 3 discontinued and 1 sample was not eligible for analysis.
  Sensitivity of the qVOA was low; 2/3 of all measurements were under the limit of detection. 6 subjects had quantifiable viral outgrowth on baseline, 8 had viral outgrowth after immunization (Day 105) and 6 had viral outgrowth after romidepsin (Day 161).
Measure: Mean (95% Confidence Interval); unit: Estimated % change from baseline
Arm/Group | Part B
Number analyzed (Participants) | 16
Estimated % change from baseline
  Total HIV-1 DNA, day 161 | -39.71 [-58.94 to -11.47]
  Integrated HIV-1 DNA, day 175 | -19.21 [-38.61 to 6.31]
  Replication competent provirus, day 161: number analyzed (Participants) | 6
  Replication competent provirus, day 161 | -38 [-67 to -8]

3. Secondary Outcome: Part A: Changes From Baseline in HIV-1 Reservoir (Total HIV-1DNA; Integrated HIV-1 DNA in Unfractionated CD4+ T Cells and Replication Competent Provirus. Estimates of Change From Baseline of the Size of the Latent HIV-1 Reservoir in CD4+ Cells.
Description: Total HIV-1 DNA and integrated HIV-1 DNA were analysed by MMRM analysis (copies/10^6 CD4+ T cells). To estimate the frequency of infectious units per 10^6 resting memory CD4+ T cells a quantitative viral outgrowth assay (qVOA) was used.
  Total HIV-1 DNA was measured at Day 84
Time Frame: Day 56/84
Population: 1 patient did not have a quantifiable load of total HIV-1 DNA at Day 84 and 2 patients diod not have a quantifiable load of replication competent provirus at day 56.
Measure: Mean (Standard Deviation); unit: copies/10^6 CD4+ T cells
Arm/Group | Part A
Number analyzed (Participants) | 6
copies/10^6 CD4+ T cells
  Total HIV-1 DNA, Basline | 791.7 (790.6)
  Total HIV-1 DNA, Day 84: number analyzed (Participants) | 5
  Total HIV-1 DNA, Day 84 | 718.8 (530.2)
  Integrated HIV-1 DNA, Baseline | 2825.6 (1145.6)
  Integrated HIV-1 DNA, Day 84 | 4846.9 (3698.4)
  Replication competent provirus, Baseline: number analyzed (Participants) | 4
  Replication competent provirus, Baseline | 0.39 (0.26)
  Replication competent provirus, Day 56: number analyzed (Participants) | 4
  Replication competent provirus, Day 56 | 0.43 (0.31)

4. Secondary Outcome: Part B: Number of Participants With Adverse Events (AE) and Serious Adverse Events (SAE)
Description: Safety and tolerability evaluation of romidepsin and Vacc-4x in combination with GM-CSF as measured by adverse events (AE) and serious adverse events (SAE).
Time Frame: 287 days
Measure: Number; unit: participants
Arm/Group | Part B
Number analyzed (Participants) | 20
participants
  Non-treatment emergent adverse events | 1
  Treatment emergent adverse events | 20
  Serious adverse event | 1
  Adverse reaction, grade 1 | 20
  Adverse reaction, grade 2 | 5
  Adverse reaction, grade 3 | 1
  Related to Vacc-4x and GM-CSF | 19
  Related to Romidepsin | 17
  Not related | 16

5. Secondary Outcome: Part B: Level of HIV-1 Transcription.
Description: At day 105, 112 and 119 patients receive romidepsin and 4 hours after each administration HIV transcription is measured as unspliced HIV-1 RNA.
Time Frame: Day 105, 112 and 119
Population: All available samples were included in this analysis; 3 withdrew consent and 2 (3 for day 119) did not have analyzable samples.
Measure: Mean (Standard Deviation); unit: copies/10^6 CD4+ T cells
Arm/Group | Part B
Number analyzed (Participants) | 15
copies/10^6 CD4+ T cells
  Day 105, before romidepsin | 6.95 (5.29)
  Day 105, 4 hours post romidepsin | 12.77 (11.19)
  Day 112, 4 hours post romidepsin | 22.98 (16.58)
  Day 119, 4 hours post romidepsin: number analyzed (Participants) | 14
  Day 119, 4 hours post romidepsin | 25.91 (21.78)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first treatment (Day 0) to the last visit (day 11 for Part A and day 287 for part B). Any signs or symptoms occurring between Screening/Visit 1 and Visit 2 (day 0)was recorded as Medical History.
Groups:
- Part B: Pre-treatment phase of 2-4 weeks (Visit 1-Visit 2) followed by a therapeutic HIV-1 immunization phase of 12 weeks (Visit 2 to Visit 7) in which 1.2 mg Vacc-4x was administered together with 0.06 mg rhuGM-CSF at Visits 2, 3, 4, 5, 6 and 7 follow by a follow-up period of 2 weeks (Visit 8).
  A viral reactivation phase of 3 weeks (Visit 9-Visit 11) consisting of one cycle of romidepsin infusion (5 mg/m2) followed by a post-treatment observation phase of ~9 weeks (Visit 12-Visit 13) to assess the effect of the investigational treatment on the size of the latent HIV-1 reservoir.
  A monitored antiretroviral pause of up to 16 weeks (Visit 14-Visit 33).
Arm/Group | Part A | Part B
Serious Adverse Events (participants affected / at risk) | 0/6 | 1/20
Other Adverse Events (participants affected / at risk) | 6/6 | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A (N=6) | Part B (N=20)
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 (0) | 1 (3) — One subject (01-225) presented three SAEs; all three were described as "alcohol withdrawal syndrome" and assessed as not related to Vacc-4x and GM-CSF and romidepsin
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A (N=6) | Part B (N=20)
Nausea (Gastrointestinal disorders) | 4 (11) | 15 (26)
Gastrointestinal sounds abnormal (General disorders) | 3 (4) | 1 (1)
Abdominal Pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (2)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 3 (5) | 15 (28)
Asthenia (General disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 4 (4)
Malaise (General disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 3 (3)
Burning sensation (Nervous system disorders) | 1 (2) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0)
Head Discomfort (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 4 (4)
Parosmia (Nervous system disorders) | 1 (1) | 1 (1)
Palpitations (Cardiac disorders) | 1 (2) | 0 (0)
Wrist Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Injection site Pruritus (General disorders) | 0 (0) | 14 (17)
Injection site erythema (General disorders) | 0 (0) | 8 (8)
Injection site pain (General disorders) | 0 (0) | 2 (2)
Feeling hot (General disorders) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 0 (0) | 1 (1)
Vomitting (Gastrointestinal disorders) | 0 (0) | 2 (3)
Colitis ulcerative (General disorders) | 0 (0) | 1 (1)
Fungal infection (Infections and infestations) | 0 (0) | 2 (2)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Parynchia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Petit mal epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Sensory disturbance (Nervous system disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Bone fissure (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Serum ferritin descreased (Investigations) | 0 (0) | 1 (1)
Viral load increased (Investigations) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Urethral discharge (Renal and urinary disorders) | 0 (0) | 1 (1)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Wisdom teeth removal (Surgical and medical procedures) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor (or designee) will prepare a final report on the study. The Investigator may not publish or present any information on this study without the express written approval of the Sponsor. Additionally, the Sponsor, may, for any reason, withhold approval for publication or presentation.